CLINICAL TRIAL: NCT06430242
Title: Role of Tele-rehabilitation in Elderly Women With Locomotor Disabilities Due to Knee Osteo Arthritis
Brief Title: Tele-rehabilitation in Knee Osteo Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prince Sattam Bin Abdulaziz University (Other)
Responsible Party: Principal Investigator, Gopal Nambi, Professor, Prince Sattam Bin Abdulaziz University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RHPT-01
Record Dates: First submitted 2024-04-28; First posted 2024-05-28 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Knee Osteoarthritis
Keywords: Knee; Osteoarthritis; Locomotor; Disability; Female
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Telerehabilitation; Exercise

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): In the active group, one of the co-investigators will install and demonstrate the use of the mobile app (Rehab App) on participants' mobile phone and explain the use of the software. The participants will be followed up for the duration of their enrolment in the e-health and tele-rehabilitation service, which can last up to 2 months and the treatment will be monitored.
  Interventions: Device: Tele rehabilitation
- Group B (Active Comparator): Participants in the control group will get the usual treatment from the clinical staff and in-person education, and they will be supervised by one of the assigned research team members every week.
  Interventions: Other: Exercise

INTERVENTIONS:
Device: Tele rehabilitation — In the active group, one of the co-investigators will install and demonstrate the use of the mobile app (Rehab App) on participants' mobile phone and explain the use of the software. The participants will be followed up for the duration of their enrolment in the e-health and tele-rehabilitation service, which can last up to 2 months.
  Arms: Group A
Other: Exercise — Participants in the control group will get the usual treatment from the clinical staff and in-person education, and they will be supervised by one of the assigned research team members every week.
  Arms: Group B

SUMMARY:
Osteoarthritis (OA) is the most common degenerative joint disease with an inflammatory component that starts from the matrix of the articular cartilage. Females are affected more than males and they have marked locomotor disabilities. Moreover, OA patients suffer from a range of extra-articular symptoms which also leads to functional impairment and disability such as fatigue, depression, anxiety, fear of movement, physical inactivity, and decreased muscle strength. OA management with physical therapy and exercise is recognized as the cornerstone of conservative and self-treatment for this chronic disease. The concept of telerehabilitation has been introduced in the field of physical medicine and rehabilitation, which combines telemedicine and rehabilitation interventions to support ongoing rehabilitation services for patients.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is the most common degenerative joint disease with an inflammatory component that starts from the matrix of the articular cartilage, progresses with disruption of chondrocyte responses and results in tissue destruction. In OA, primary involvement is seen in the articular cartilage, and progressive damage occurs. Females are affected more than males and they have marked locomotor disabilities. Moreover, OA patients suffer from a range of extra-articular symptoms which also leads to functional impairment and disability such as fatigue, depression, anxiety, fear of movement, physical inactivity, and decreased muscle strength.

OA management with physical therapy and exercise is recognized as the cornerstone of conservative and self-treatment for this chronic disease. The lack of professional supervision and feedback will result in reduced participation in continuing OA medical or rehabilitative services, which in turn will reduce the effectiveness of OA treatments.

With the development of telemedicine, it has been determined that patients living in remote areas have the chance to communicate with professional physicians simultaneously. The concept of telerehabilitation has been introduced in the field of physical medicine and rehabilitation, which combines telemedicine and rehabilitation interventions to support ongoing rehabilitation services for patients. Internet- based rehabilitation is one of the effective strategies in telerehabilitation. The use of the internet to provide health-related interventions has the potential to reduce the cost of treatment and improve user satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with mild to moderate OA by their physicians.
* Female in the age range of 45 - 65 years.
* Volunteer to participate in the study.
* Living independently.
* Being able to walk without using an assistive device.
* Owning a mobile phone, tablet, or computer with an internet connection.
* Being able to use the device without assistance.

Exclusion Criteria:

* Having been diagnosed with any other systemic rheumatic diseases.
* Having been involved in a physiotherapy and rehabilitation program in any health institution in the last 6 months,
* Having knee-related surgery,
* Having meniscal or ligament-associated tears occurred in the past 6 months,
* Having a history of falling more than 2 times in the last 6 months,
* Having a history of knee injection in the last 4 weeks or scheduled in the next 8 week,
* Being illiterate, having cognitive problems, having blurred vision problem, and having hearing loss.

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female participants in the age range of 45 - 65 years.
Enrollment: 56 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-04-20 (Actual); Study Completion 2024-04-20 (Actual)

PRIMARY OUTCOMES:
Pain intensity | Baseline
  Which was measured by 10 cm visual analogue scale
Pain intensity | 2 months
  Which was measured by 10 cm visual analogue scale
Pain intensity | After 6 months
  Which was measured by 10 cm visual analogue scale

SECONDARY OUTCOMES:
Functional disability | Baseline
  Which was measured by WOMAC questionnaire
Functional disability | 2 months
  Which was measured by WOMAC questionnaire
Functional disability | 6 months
  Which was measured by WOMAC questionnaire
Gait velocity | Baseline
  Which was measured in meters/ second
Gait velocity | 2 months
  Which was measured in meters/ second
Gait velocity | 6 months
  Which was measured in meters/ second
Step length | Baseline
  Which was measured in meters
Step length | 2 months
  Which was measured in meters
Step length | 6 months
  Which was measured in meters
Cadence | Baseline
  Which was measured in number of steps per minute
Cadence | 2 months
  Which was measured in number of steps per minute
Cadence | 6 months
  Which was measured in number of steps per minute
Quality | Baseline
  Which was measured with KOOS questionnaire
Quality | 2 months
  Which was measured with KOOS questionnaire
Quality | 6 months
  Which was measured with KOOS questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Gopal Nambi, Al Kharj, Riyadh Region, Saudi Arabia